CLINICAL TRIAL: NCT05511766
Title: The Potential Role of Allopurinol Versus Atorvastatin to Prevent Complications of Liver Cirrhosis: A Quadruple Blind Clinical Study
Brief Title: Allopurinol Versus Atorvastatin to Prevent Complications of Liver Cirrhosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Khadija Ahmed Mhrose Glal, Assistant lecturer of clinical pharmacy- Clinical pharmacy department- Faculty of pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: allopurinol v atorvastatin
Record Dates: First submitted 2022-08-17; First posted 2022-08-23 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Cirrhosis; Hepatic Encephalopathy; Ascites; Varices; SBP - Spontaneous Bacterial Peritonitis
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy; Ascites; Varicose Veins | interventions — Allopurinol; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PLACEBO (Placebo Comparator): Group1: (Placebo, n=50) who will receive oral placebo tablet once daily FOR 6 MONTHS
  Interventions: Drug: Placebo
- Allopurinol (Active Comparator): Group 2:(Allopurinol n=50) who will receive oral allopurinol 300 mg daily for 6 months
  Interventions: Drug: Allopurinol 300 MG
- Simvastatin (Active Comparator): Group 3: (atorvastatin n=50) who will receive oral atorvastatin 20 mg daily for 6 months
  Interventions: Drug: Atorvastatin 20mg

INTERVENTIONS:
Drug: Allopurinol 300 MG — a competitive xanthine oxidase inhibitor, reduces oxidative stress and attenuates bacterial translocation
  Other Names: zyloric
  Arms: Allopurinol
Drug: Atorvastatin 20mg — is lipid-lowering agent with anti-oxidative stress and anti-inflammation properties
  Arms: Simvastatin
Drug: Placebo — not containing drugs
  Arms: PLACEBO

SUMMARY:
The study aims to compare the potential benefit of allopurinol versus atorvastatin in reducing the risk of developing cirrhosis-related complications, delaying the onset of hepatocellular carcinoma, and improving survival. Furthermore, the study aims to evaluate their impact on parents' related quality of life.

DETAILED DESCRIPTION:
Cirrhosis is the late stage of liver damage and possess two phases: a compensated phase with favorable prognosis and a decompensated phase with high mortality rate1.The shift from compensated to decompensated cirrhosis is characterized by the onset of complications, including ascites, hepatic encephalopathy (HE), variceal bleeding, and spontaneous bacterial peritonitis (SBP) which are associated with substantial morbidity and negative Impact on quality of life (QOL)2.

The gut microbiota plays an important role in cirrhosis and development of cirrhosis-related complications3.

Indeed, translocation of endotoxins is increased in patients with cirrhosis and patients with more severe cirrhosis (i.e. Patients with decompensated cirrhosis, hospitalized patients) had significantly greater serum endotoxin concentrations that mediate complications of cirrhosis4.

Intestinal permeability plays a role in the development of bacterial translocation and may be involved in the development of complications of cirrhosis5. This 'leaky gut' phenomenon increases with the degree of liver failure and is particularly prominent in patients with cirrhosis who have experienced severe septic complications and has been implicated in the hepatic production of endotoxin-associated proinflammatory cytokines6.

Intestinal mucosa alterations at the subcellular level have been reported in experimental cirrhosis, in relation to an increased oxidative stress due to overactivity in the enzyme xanthine oxidase7.

Allopurinol, a competitive xanthine oxidase inhibitor, reduces oxidative stress and attenuates bacterial translocation in portal hypertensive animals, suggesting that the damaging effects of oxygen-derived free radicals and peroxidation on mucosal cells may be counteracted by a free radical scavenger8.

In 2007, a pilot study demonstrated that allopurinol in patients with cirrhosis is associated with a significant reduction in oxidative stress but no effect on intestinal permeability and inflammatory markers. The study duration was only 10 days and therefore another study with a long period of time is essential 9.

Statins are one class of medications being studied to determine their effect on progression and decompensation of CLDs. Besides their lipid-lowering effects, statins also decrease oxidative stress and inflammation by decreasing activation of inflammatory cells, and improve endothelial function by increasing synthesis of nitric oxide, restoring the function of endothelial cells, and increasing the number of endothelial progenitors cells10. Recent studies have suggested an association between statin use and hepatic decompensation in patients with CLDs11.

Cirrhosis and its complications have a substantial economic, social, and personal impact on affected patients, as well as their families and caregivers12. Given that the number of primary prophylaxis treatments that prevent complications of cirrhosis is limited. Therefore, it is important to examine whether allopurinol and statins have the potential to reduce the risk of developing several complications of cirrhosis, including HE, SBP, variceal bleeding, hepatocellular carcinoma (HCC) and hepatorenal syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria
* Age 18 to 75 years old
* Both sex
* Adults with cirrhosis in a stable conditions

Exclusion Criteria:

* Exclusion criteria
* Active SBP
* Renal insufficiency (serum creatinine > 2.0 mg/dl)
* Active GIT hemorrhage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-04-25 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of breakthrough episodes of cirrhosis related complication during treatment | 6 months
  Number of breakthrough episodes of cirrhosis related complication during 6 month

CONTACTS AND LOCATIONS:
Overall Officials: khadija glal, Principal Investigator — assistant lecturer
Locations (1):
- Tanta University, Tanta, Egypt